CLINICAL TRIAL: NCT07234448
Title: Evaluation of the Use of a Probiotic Containing Bifidobacterium Breve PRL2020 in Oral Drops in Preventing Side Effects From Amoxicillin or Amoxicillin/Clavulanic Acid Antibiotic Use: a Multicentre, Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Evaluation of the Use of a Probiotic Containing Bifidobacterium Breve PRL2020 in Oral Drops in Preventing Side Effects From Amoxicillin or Amoxicillin/Clavulanic Acid Antibiotic Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Brevicillin_PRL2020_Trial
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Antibiotic-associated Diarrhea

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to receive either Brevicillin® gocce containing Bifidobacterium breve PRL2020 or a matching placebo, both administered only during the antibiotic treatment period (6-10 days, according to physician prescription). After completion of antibiotic therapy, all participants enter a follow-up period through day 15 without probiotic or placebo administration.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design: both participants, care providers, investigators, and outcome assessors are unaware of treatment assignments. The probiotic and placebo products are identical in appearance, packaging, and labeling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brevicillin® gocce (Bifidobacterium breve PRL2020) (Experimental): Participants will receive Brevicillin® gocce, a probiotic food supplement containing Bifidobacterium breve PRL2020 (LMG S-32458), alongside standard antibiotic therapy with amoxicillin or amoxicillin/clavulanic acid.
  Dosage and administration: 5 drops, 2-3 times per day (depending on antibiotic dosing schedule), administered during the antibiotic treatment period (6-10 days). After completion of antibiotic therapy, participants will enter a follow-up period until day 15 without probiotic administration.
  Interventions: Dietary Supplement: Brevicillin® gocce (Bifidobacterium breve PRL2020)
- Placebo (Placebo Comparator): Participants will receive a placebo formulation matched in appearance, packaging, and dosing schedule to Brevicillin® gocce, administered alongside standard antibiotic therapy with amoxicillin or amoxicillin/clavulanic acid.
  The placebo will be given at the same frequency (5 drops, 2-3 times per day) and duration as the experimental product during the antibiotic treatment period (6-10 days). After antibiotic completion, participants will enter a follow-up period until day 15 without placebo administration.
  Interventions: Other: Placebo (matching oil drops)

INTERVENTIONS:
Dietary Supplement: Brevicillin® gocce (Bifidobacterium breve PRL2020) — Brevicillin® gocce is a probiotic dietary supplement in oily drops containing the bacterial strain Bifidobacterium breve PRL2020 (LMG S-32458). Each 5-drop dose contains approximately 5 billion live cells. The supplement is administered orally 2-3 times per day, in parallel with antibiotic therapy (amoxicillin or amoxicillin/clavulanic acid), for 6-10 days only (during the antibiotic course).
  After completion of antibiotic therapy, participants enter a follow-up period until day 15 without probiotic administration. The product is manufactured by PharmExtracta S.p.A., Pontenure, Italy.
  Arms: Brevicillin® gocce (Bifidobacterium breve PRL2020)
Other: Placebo (matching oil drops) — The placebo is a formulation identical in appearance, packaging, and administration schedule to Brevicillin® gocce but without the Bifidobacterium breve PRL2020 strain. It is administered orally 2-3 times per day only during the antibiotic treatment period (6-10 days).
  After antibiotic completion, participants enter a follow-up period until day 15 without placebo administration.
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled clinical trial will evaluate the efficacy and safety of the probiotic Bifidobacterium breve PRL2020 (Brevicillin® gocce) in preventing gastrointestinal side effects associated with antibiotic therapy using amoxicillin or amoxicillin/clavulanic acid in pediatric patients aged 0-12 years. Participants will be randomized 1:1 to receive either the probiotic supplement or placebo during standard antibiotic treatment for 6-10 days, followed by a post-treatment observation period up to day 15 without probiotic or placebo administration. The primary objective is to assess the reduction in the incidence of antibiotic-associated diarrhea (AAD).

DETAILED DESCRIPTION:
Antibiotic therapy with amoxicillin or amoxicillin/clavulanic acid is widely prescribed in pediatric populations but is frequently associated with gastrointestinal adverse effects, particularly diarrhea. These effects are linked to disruption of the gut microbiota and a reduction in bifidobacterial populations. Bifidobacterium breve PRL2020 is a probiotic strain with demonstrated intrinsic, non-transferable resistance to these antibiotics and has been developed to mitigate antibiotic-induced dysbiosis.

This study is a multicenter, prospective, randomized, double-blind, placebo-controlled, non-profit trial conducted in pediatric centers across Italy. The study aims to evaluate the clinical efficacy and safety of Bifidobacterium breve PRL2020 in reducing the incidence and severity of antibiotic-associated diarrhea (AAD) in children receiving amoxicillin or amoxicillin/clavulanic acid.

A total of 1,000 participants (500 per group) will be enrolled. Participants will be randomized 1:1 to receive either Brevicillin® gocce (5 drops 2-3 times daily, containing 5 billion CFU of B. breve PRL2020 per dose) or matching placebo only during antibiotic therapy (6-10 days). After completion of antibiotic treatment, participants will enter a follow-up period until day 15 without probiotic or placebo administration.

The primary outcome is the incidence of AAD, defined as ≥3 diarrheal episodes in one day during antibiotic treatment (Bristol Stool Scale 5-7).

Secondary outcomes include the incidence and duration of diarrhea, daily bowel movements, stool consistency, gastrointestinal and extra-intestinal symptoms (such as nausea, vomiting, abdominal pain), treatment compliance, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 0-12 years.
* Undergoing antibiotic therapy with amoxicillin or amoxicillin/clavulanic acid.
* Parent or legal guardian provides written informed consent.

Exclusion Criteria:

* Use of antibiotic therapy within 4 weeks prior to enrolment.
* Use of other probiotic products or lactic acid bacteria during the study.
* Pre-existing diarrhea within 4 weeks prior to enrolment.
* Chronic inflammatory bowel disease.
* Immunodeficiency.
* Lack of parental or legal guardian consent to participate in the study.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Antibiotic-Associated Diarrhea (AAD) | 15 days
  Evaluation of the efficacy of Bifidobacterium breve PRL2020 (Brevicillin® gocce) in reducing the incidence of antibiotic-associated diarrhea (AAD), defined as ≥3 diarrheal episodes within one day of antibiotic treatment, with stool consistency corresponding to types 5-7 on the Bristol Stool Scale. Data will be collected through a daily diary completed by the parent or legal guardian.

SECONDARY OUTCOMES:
Incidence of children with at least one episode of diarrhea | 15 days
  Number of participants experiencing at least one episode of diarrhea during the study period, as recorded in the daily diary.
Number of daily defecations | 15 days
  Average number of daily bowel movements recorded by the parent or guardian during the study period, using the child's daily diary.
Number of days with diarrhea | 15 days
  Total number of days in which diarrhea occurs during the observation period, recorded by the parent or guardian.
Stool consistency | 15 days
  Assessment of stool consistency using the Bristol Stool Scale (BSS) to evaluate changes in bowel habits during and after antibiotic treatment.
Gastrointestinal and extra-intestinal symptoms | 15 days
  Evaluation of symptoms related to antibiotic use, including abdominal pain, nausea, and vomiting, assessed from daily diary entries completed by the parent or guardian
Treatment compliance | 15 days
  Assessment of adherence to the probiotic or placebo regimen, graded by the pediatrician on a scale from "poor" to "excellent" at the end of the study period.
Adverse events | 15 days
  Documentation and evaluation of any adverse events reported during treatment and follow-up, as recorded in the child's daily diary and verified by the study physician.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Sisti, PhD, Principal Investigator — University of Urbino "Carlo Bo"

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bartlett JG. Clinical practice. Antibiotic-associated diarrhea. N Engl J Med. 2002 Jan 31;346(5):334-9. doi: 10.1056/NEJMcp011603. No abstract available. PMID 11821511
- [Background] Salvo F, Polimeni G, Moretti U, Conforti A, Leone R, Leoni O, Motola D, Dusi G, Caputi AP. Adverse drug reactions related to amoxicillin alone and in association with clavulanic acid: data from spontaneous reporting in Italy. J Antimicrob Chemother. 2007 Jul;60(1):121-6. doi: 10.1093/jac/dkm111. Epub 2007 Apr 21. PMID 17449881
- [Background] Caron F, Ducrotte P, Lerebours E, Colin R, Humbert G, Denis P. Effects of amoxicillin-clavulanate combination on the motility of the small intestine in human beings. Antimicrob Agents Chemother. 1991 Jun;35(6):1085-8. doi: 10.1128/AAC.35.6.1085. PMID 1929247
- [Background] Yang L, Bajinka O, Jarju PO, Tan Y, Taal AM, Ozdemir G. The varying effects of antibiotics on gut microbiota. AMB Express. 2021 Aug 16;11(1):116. doi: 10.1186/s13568-021-01274-w. PMID 34398323
- [Background] Mancabelli L, Mancino W, Lugli GA, Argentini C, Longhi G, Milani C, Viappiani A, Anzalone R, Bernasconi S, van Sinderen D, Ventura M, Turroni F. Amoxicillin-Clavulanic Acid Resistance in the Genus Bifidobacterium. Appl Environ Microbiol. 2021 Mar 11;87(7):e03137-20. doi: 10.1128/AEM.03137-20. Print 2021 Mar 11. PMID 33483308
- [Background] Di Pierro F, Campedelli I, De Marta P, Fracchetti F, Del Casale A, Cavecchia I, Matera M, Cazzaniga M, Bertuccioli A, Guasti L, Zerbinati N. Bifidobacterium breve PRL2020: Antibiotic-Resistant Profile and Genomic Detection of Antibiotic Resistance Determinants. Microorganisms. 2023 Jun 24;11(7):1649. doi: 10.3390/microorganisms11071649. PMID 37512822
- [Background] Biasucci G, Capra ME, Giudice A, Monopoli D, Stanyevic B, Rotondo R, Mucci A, Neglia C, Campana B, Esposito S. Use of Probiotics During Antibiotic Therapy in Pediatrics: A Cross-Sectional Survey of Italian Primary Care Pediatricians. Antibiotics (Basel). 2025 Jun 4;14(6):577. doi: 10.3390/antibiotics14060577. PMID 40558167